CLINICAL TRIAL: NCT07090070
Title: Evaluating Treatment Strategies for p53 Mutant Oral Epithelial Dysplasia and SCC Study
Brief Title: Evaluating Treatment Strategies for p53 Mutant Oral Cancer and Oral Cancer Precursors: A Randomized Controlled Trial
Acronym: p53 RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Eitan Prisman, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H25-01056
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Oral Epithelial Dysplasia (OED); Oral Squamous Cell Carcinoma (SCC)
Keywords: p53 mutant; SCC; oral epithelial dysplasia
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Endoglin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1: p53 mutant mild/moderate dysplasia observational group (No Intervention): Observation only
- Cohort 1: p53 mutant mild/moderate dysplasia excision group (Experimental): Clear margin excision of the lesion under local anesthetic, with re-excision for p53-positive margins
  Interventions: Procedure: Cohort 1 Intervention group
- Cohort 2: p53 mutant Severe/CIS dysplasia clear severe/CIS margin group (Active Comparator): Clear margin excision of the lesion under local anesthetic, with re-excision until severe/CIS margins are clear
  Interventions: Procedure: Cohort 2 severe/CIS margins clear
- Cohort 2: p53 mutant Severe/CIS dysplasia negative p53 and severe/CIS margin group (Experimental): Excision of the lesion ensuring final negative p53 and severe/CIS margins
  Interventions: Procedure: Cohort 2 p53 and severe/CIS margins clear
- Cohort 3: p53 mutant T1 SCC (DOI 0-3mm) excision and END group (Active Comparator): Excision of primary lesion with 5+ mm margins and immediate elective neck dissection (END)
  Interventions: Procedure: Cohort 3 Excision and END
- Cohort 3: p53 mutant T1 SCC (DOI 0-3mm) excision and follow up group (Experimental): Excision of primary lesion with 5+mm margins and close follow up with salvage elective neck dissection (END) if development of nodal disease
  Interventions: Procedure: Cohort 3 Excision and Close follow up

INTERVENTIONS:
Procedure: Cohort 1 Intervention group — Clear margin excision of the lesion under local anesthetic, with re-excision for p53-positive margins.
  Arms: Cohort 1: p53 mutant mild/moderate dysplasia excision group
Procedure: Cohort 2 severe/CIS margins clear — Clear margin excision of the lesion under local anesthetic, with re-excision until severe/CIS margins are clear
  Arms: Cohort 2: p53 mutant Severe/CIS dysplasia clear severe/CIS margin group
Procedure: Cohort 2 p53 and severe/CIS margins clear — Excision of the lesion ensuring final negative p53 and severe/CIS margins
  Arms: Cohort 2: p53 mutant Severe/CIS dysplasia negative p53 and severe/CIS margin group
Procedure: Cohort 3 Excision and END — Excision of primary lesions with 5+mm margins and immediate elective neck dissection
  Arms: Cohort 3: p53 mutant T1 SCC (DOI 0-3mm) excision and END group
Procedure: Cohort 3 Excision and Close follow up — Excision of primary lesion with 5+mm margins and close follow up with salvage elective neck dissection if development of nodal disease
  Arms: Cohort 3: p53 mutant T1 SCC (DOI 0-3mm) excision and follow up group

SUMMARY:
The goal of this clinical trial is to optimize treatment strategies for patients with p53-mutant oral epithelial dysplasia (OED) and early-stage oral squamous cell carcinoma (SCC). The main question it aims to answer is what the most optimal treatment is at each diagnostic stage. It is hypothesized that lesions with p53-abnormal low-grade dysplasia without surgical intervention will progress to high-grade dysplasia or SCC in 4 years. It is also predicted that a clear p53 and severe/CIS excision margins in patients with p53-abnormal HGD will reduce the progression to invasive SCC, compared to clear severe/CIS margins, within 4 years. Finally, it is thought that patients with p53-abnormal cT1N0 and DOI<3mm receiving an END will have improved disease free and overall survival. This research will elucidate whether or not these hypotheses are correct.

Participants in each diagnostic cohort will be assigned to one of two different treatment options, listed below:

Cohort 1:

A) No intervention, observation only B) Surgical excision with clear margins

Cohort 2:

A) Surgical excision with clear severe/CIS margins B) Surgical excision with clear severe/CIS and p53 margins

Cohort 3:

A) Surgical excision and elective neck dissection (END) B) Surgical excision and close follow-up, only END if development of nodal disease

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or over

Cohort 1:

* Biopsy-confirmed mild/moderate dysplasia with p53 mutations (tested via IHC)
* No prior treatment for oral premalignant lesions
* No clinical evidence of SCC

Cohort 2:

* Biopsy-confirmed severe dysplasia or CIS with p53 mutation (tested via IHC)

Cohort 3:

* T1 SCC with p53 mutation (tested via IHC)
* Depth of Invasion (DOI) 0-3mm
* Clinically and radiologically node-negative (confirmed by contrast-enhanced CT)

Exclusion Criteria:

* History of head and neck radiation
* Immunocompromised status
* Location of excision would be functionally morbid
* Lesions greater than 3cm
* Presence of Proliferative Verrucous Leukoplakia

Cohort 1:

* Severe dysplasia or carcinoma is situ (CIS) on initial biopsy

Cohort 2:

* Presence of invasive SCC on initial biopsy

Cohort 3:

* Positive nodes on imaging
* DOI >= 4mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2032-01 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Progression to severe/CIS dysplasia or SCC | 4 years
  Whether diagnosis progressed from mild/moderate OED to severe/CIS dysplasia or SCC.
Progression to invasive SCC | 4 years
  Whether diagnosis progressed from severe/CIS dysplasia to invasive SCC.
Disease free survival | 4 years
  If survival is achieved disease free following treatment.

SECONDARY OUTCOMES:
Time to progression | 4 years
  How long it took for disease diagnosis to progress
Overall survival | 4 years
  Overall survival is measured as survival for 4 years following diagnosis and treatment.
p16 status | 4 years
  p16 mutation status, as assessed by IHC using pattern-based interpretation

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] D'Cruz AK, Vaish R, Kapre N, Dandekar M, Gupta S, Hawaldar R, Agarwal JP, Pantvaidya G, Chaukar D, Deshmukh A, Kane S, Arya S, Ghosh-Laskar S, Chaturvedi P, Pai P, Nair S, Nair D, Badwe R; Head and Neck Disease Management Group. Elective versus Therapeutic Neck Dissection in Node-Negative Oral Cancer. N Engl J Med. 2015 Aug 6;373(6):521-9. doi: 10.1056/NEJMoa1506007. Epub 2015 May 31. PMID 26027881
- [Background] Liu KY, Durham JS, Wu J, Anderson DW, Prisman E, Poh CF. Nodal Disease Burden for Early-Stage Oral Cancer. JAMA Otolaryngol Head Neck Surg. 2016 Nov 1;142(11):1111-1119. doi: 10.1001/jamaoto.2016.2241. PMID 27560665
- [Background] Durham JS, Brasher P, Anderson DW, Yoo J, Hart R, Dort JC, Seikaly H, Kerr P, Rosin MP, Poh CF. Effect of Fluorescence Visualization-Guided Surgery on Local Recurrence of Oral Squamous Cell Carcinoma: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2020 Dec 1;146(12):1149-1155. doi: 10.1001/jamaoto.2020.3147. PMID 33034628
- [Background] Hyodo T, Kuribayashi N, Fukumoto C, Komiyama Y, Shiraishi R, Kamimura R, Sawatani Y, Yaguchi E, Hasegawa T, Izumi S, Wakui T, Nakashiro KI, Uchida D, Kawamata H. The mutational spectrum in whole exon of p53 in oral squamous cell carcinoma and its clinical implications. Sci Rep. 2022 Dec 15;12(1):21695. doi: 10.1038/s41598-022-25744-8. PMID 36522371
- [Background] Lin TY, Liu KYP, Novack R, Mattu PS, Ng TL, Hoang LN, Prisman E, Poh CF, Ko YCK. Abnormal p53 Immunohistochemical Patterns Are Associated with Regional Lymph Node Metastasis in Oral Cavity Squamous Cell Carcinoma at Time of Surgery. Mod Pathol. 2024 Dec;37(12):100614. doi: 10.1016/j.modpat.2024.100614. Epub 2024 Sep 10. PMID 39265952
- [Background] Gleber-Netto FO, Neskey D, Costa AFM, Kataria P, Rao X, Wang J, Kowalski LP, Pickering CR, Dias-Neto E, Myers JN. Functionally impactful TP53 mutations are associated with increased risk of extranodal extension in clinically advanced oral squamous cell carcinoma. Cancer. 2020 Oct 15;126(20):4498-4510. doi: 10.1002/cncr.33101. Epub 2020 Aug 14. PMID 32797678
- [Background] Liu KYP, Zhu SY, Harrison A, Chen ZY, Guillaud M, Poh CF. Quantitative nuclear phenotype signatures predict nodal disease in oral squamous cell carcinoma. PLoS One. 2021 Nov 4;16(11):e0259529. doi: 10.1371/journal.pone.0259529. eCollection 2021. PMID 34735529
- [Background] Novack R, Zhang L, Hoang LN, Kadhim M, Ng TL, Poh CF, Kevin Ko YC. Abnormal p53 Immunohistochemical Patterns Shed Light on the Aggressiveness of Oral Epithelial Dysplasia. Mod Pathol. 2023 Jul;36(7):100153. doi: 10.1016/j.modpat.2023.100153. Epub 2023 Mar 9. PMID 36906072
- [Background] Ko YCK, Liu KYP, Chen E, Zhu SY, Poh CF. p53 Abnormal Oral Epithelial Dysplasias are Associated With High Risks of Progression and Local Recurrence-A Retrospective Study in a Longitudinal Cohort. Mod Pathol. 2024 Dec;37(12):100613. doi: 10.1016/j.modpat.2024.100613. Epub 2024 Sep 10. PMID 39265950